CLINICAL TRIAL: NCT02708940
Title: Participatory Messaging in the UCLA Psychiatry Partial Hospitalization and Intensive Outpatient Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#14-001879
Record Dates: First submitted 2016-02-04; First posted 2016-03-15 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Depression; Anxiety; Psychosis
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Control arm - these patients will get usual care as part of the PHP and IOP programs at UCLA. They will not receive mobile support messages.
  Interventions: Other: Usual Care
- Participatory technology development (Active Comparator): Intervention - Patients will have access to a website that allows them to co-create mobile support messages with their therapist to support their care as part of the PHP and IOP programs at UCLA.
  Interventions: Other: Participatory technology development

INTERVENTIONS:
Other: Participatory technology development — Creating mobile support tools by patients and their therapists
  Arms: Participatory technology development
Other: Usual Care — Usual care as part of the UCLA PHP and IOP programs
  Arms: Usual care

SUMMARY:
This research project aims to evaluate the feasibility and effectiveness of a new approach to tailored mobile applications using the Chorus Participatory Mobile Framework. PHP and IOP program participants-patients and therapists--will be consented and enrolled by study staff. Study participants will be invited to workgroups specific to their program to discuss the usability of Chorus and be asked to complete surveys on demographics, satisfaction, self-efficacy, and involvement with Chorus and usability of the tool.

DETAILED DESCRIPTION:
The Partial Hospitalization Program (PHP) and Intensive Outpatient Program (IOP) in the Neuropsychatric Hospital at UCLA provide psychiatric services for adults and children with acute mental illness. These include voluntary programs that support individuals in their recovery with the goal to assist patients in achieving the highest level of independence. Most programs operate Monday through Friday between four to eight hours a day. Recently, the PHP and IOP programs have decided to start including mobile messaging as a part of care, helping patients to feel supported even after they have left the hospital for the day.

The purpose of this study is to evaluate the feasibility and effectiveness of their ongoing use of the Chorus Participatory Mobile Framework to support clinical care. Chorus is a framework and web application that allows users to rapidly create a broad range of automated text messaging (SMS), interactive voice (IVR), or mobile web applications using a simple and accessible visual interface without requiring any server programming. There will be two broad populations using Chorus: (1) programs (e.g. OCD Intensive Treatment Program) in which all participants will receive participatory mobile messaging and (2) programs (e.g. Adult Acute PHP) in which patients will be randomized to receive either participatory mobile messaging or no mobile messaging. Across all programs, Kandace Whiting and Armen Arevian will train PHP and IOP therapists starting with creating simple, basic, useful messaging content in Chorus to support patients in achieving program goals. Examples of messages include Cognitive Behavioral Therapy (CBT), symptom management, and stress management cues to patients in the Obsessive Compulsive Disorder Clinic, patients in the Adult Eating Disorder Clinic, and parents from The Achievement, Behavior, Cognition (ABC) Child Programs.

All participating patients receiving participatory mobile messaging will work with program staff one-on-one to tailor SMS and IVR content and design based on their own preferences. By being able to personalize the messaging, the Chorus Participatory Mobile Framework meets the capacities and preferences of the users rather than a "one-size" approach requiring adaptation of the users to the technology. Both therapists and patients will be invited to up to bi-weekly, in-person workshops specific to their program to provide feedback and input. The goal of these workshops is to further develop and refine the novel mobile interventions based on stakeholder input. The Chorus Participatory Framework will be used during the workshops to develop and test the application in real-time. Workshops will be audio and/or video recorded to document the process.

ELIGIBILITY:
Inclusion Criteria:

* Patients (over the age of 18) or parents of patients who are minors (between the ages of 6 and 17)
* Enrolled in PHP or IOP programs at Resnick Neuropsychiatric Hospital
* Agree to participate (minors will be required to have parental consent)
* Patient participants will need to be English speaking because text and IVR messages and workshops will be conducted in English.
* Patient must have cellular phone that can receive text messages
* All PHP and IOP staff are eligible and will be invited to participate in workshops and complete surveys.

Exclusion Criteria:

* Declines consent or is unwilling to participate in the study
* Does not speak English. Language other than English is an exclusion given resources and capacity of the study
* Patients without a cellular phone that can receive text messages
* Not receiving texts or IVR messages from their program is an exclusion given that it is the intervention we are evaluating
* Patients under the age of 6.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in homework completion rate | Collected on each program attendance day (up to daily), through discharge from program, an average of 12 weeks
  the change in the degree to which patients complete tasks assigned to them by their provider as part of their treatment

SECONDARY OUTCOMES:
length of stay | At discharge from program, an average of 12 weeks
  length of stay (in terms of days and hours/day of program attendance)
time to discharge | From admission to program until discharge from program, assessed up to 20 weeks
  time to step down from partial hospitalization program to intensive outpatient program and time to discharge from program
Number of patient visits to health care organizations outside of clinic | at patient disenrollment from study, approximately 3 months after discharge from program, up to 40 weeks
  the number of services that patients utilize outside of the clinic, including ED visits and inpatient hospitalizations.
Types of health care services patients utilize outside of clinic | at patient disenrollment from study, approximately 3 months after discharge from program, up to 40 weeks
  the types of services that patients utilize outside of the clinic, including ED visits and inpatient hospitalizations.
change in depression symptoms | Upon admission to program, at mid-point of stay in program, at discharge from program (may also be up to weekly during stay), an average of 12 weeks; and 3 months after discharge from programa
  PHQ-9 to measure changes in depression symptoms
Change in Patient Treatment Self-Efficacy | weekly during stay in program, through discharge from program, an average of 12 weeks
  change patient treatment self-efficacy from week-to-week during program
Difference in Patient Satisfaction with Program between Intervention vs Control groups | at discharge from program, an average of 12 weeks
  comparing patient satisfaction with services and support between the intervention and control groups
Messaging Application Usability | weekly during stay in program, through discharge from program, an average of 12 weeks
  Weekly survey of patients in the intervention arm and all providers to assess the usability of the messaging application
Patient Involvement in Message Development | weekly during stay in program, through discharge from program, an average of 12 weeks
  Completed by patients in the intervention arm and by provider for each patient in intervention arm to assess the extent of patient involvement in the development of message content and schedule, and use of messaging application

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Partial Hospitalization and Intensive Outpatient Programs, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No